CLINICAL TRIAL: NCT04590352
Title: Mucosal Immunity in Patients Diagnosed With SARS-CoV-2 Infection and Their Household Contacts
Brief Title: Mucosal Immunity Against SARS-CoV-2 Infection in COVID-19 Patients
Acronym: MuCo
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-6342; NL73418.091.20 (Registry Identifier: CCMO)
Record Dates: First submitted 2020-08-27; First posted 2020-10-19 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2020-07

CONDITIONS: SARS-CoV-2 Infection
Keywords: SARS-CoV-2; household contacts; mucosal immunitiy; antibodies
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — nasopharyngeal and throat swab, mucosal lining fluid, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Index case and household contacts: * nasophryngeal and throat swab at day 0.
  * collection of mucosal lining fluid: day 0, 7, 14, 28 for index case and day 0, 3, 6, 28 for household contacts.
  * fingerprick at day 28 (optional).
  * daily record of symptoms from day 0-28.
  Interventions: Procedure: nasopharyngeal and throat swab; Procedure: collection of mucosal lining fluid; Procedure: blood collection via fingerprick

INTERVENTIONS:
Procedure: nasopharyngeal and throat swab — diagnostic specimens via nasopharyngeal swab and throat swab were collected following the current standard operating procedures.
Procedure: collection of mucosal lining fluid — MLF will be collected via nasal absorption at the inclusion visit by study staff and four more time points by the parents or by the children themselves. Nasal absorption is performed by maneuvering a strip of synthetic absorptive matrices (SAM) into the lumen of the nostril, avoiding rubbing against the nasal mucosa. The outside of the nose is then pressed with a finger to cause apposition of the SAM against the mucosa.
Procedure: blood collection via fingerprick — Participants will be asked to wash their hands with soap and warm water. The procedure involves cleaning the ball of the fingertip with an alcohol swab, then using a sterile disposable lancet to pierce the skin (BD Microtainer Lancet or similar). The lancet is placed in a spring-loaded device, which propels the lancet a fixed distance (a few mm) into the skin when the trigger is pressed. Approximately 10-20 drops of blood (0.3 ml) will then be collected with a sterile capillary tube. The participant is given a cotton wool pad to mop up any extra blood, and an elastoplast-type bandage is placed over the finger if necessary. Fingerprick blood samples will only be collected from participants older than 6 months at 28-32 days after the first home visit (d0). Lancet length will be adjusted for age (2.0 mm for participants 8 years and older, 1.5 mm for participants older than 6 months and younger than 8 years).

SUMMARY:
In this study nasal fluid (mucosal lining fluid), nose and throat swabs and blood was collected from patients with a confirmed SARS-CoV-2 infection who remained in home isolation, as well as from their household contacts who remained in home quarantine. On the collected nose and throat swabs a coronavirus PCR was performed. Antibodies against SARS-CoV-2 were measured in the mucosal lining fluid and blood samples.

DETAILED DESCRIPTION:
Objective:

Primary Objective: to analyse the development of mucosal immunity against SARS-CoV-2 in nasal fluid of Covid-19 patients and their household contacts

Secondary Objective(s):

* To descriptively analyse the correlation of mucosal antibodies with viral diagnostics and disease symptoms
* To determine the correlation between mucosal and serum antibody levels
* To study the functionality of serum and mucosal antibodies

Study design: A single-site, observational, prospective cohort study among COVID-19 patients and their household contacts Study population: The study will be conducted among COVID-19 patients with a laboratory-confirmed infection with SARS-CoV-2, as well as household contacts remaining in home quarantine at the same address, among secondary and tertiary hospital careworkers in the provinces of Gelderland and Noord-Brabant in The Netherlands.

Intervention (if applicable): N/A

Main study parameters/endpoints:

Mucosal antibodies: descriptive analysis of SARS-CoV-2 IgG, IgA, IgM and IgD concentrations in nasal fluid at the various collection moments.

Viral diagnostics: presence of SARS-CoV-2 in diagnostic specimens collected at inclusion visit.

Disease symptoms: presence of respiratory complaints in participants. Serum antibodies: descriptive analysis of SARS-CoV-antibody concentrations in serum at day 28 Antibody functionality: descriptive analysis of antibody functionality of serum and nasal fluid samples, including virus neutralization

ELIGIBILITY:
Inclusion Criteria:

* Index case:

  * Laboratory-confirmed case of SARS-CoV-2, with a positive indication for home isolation, and;
  * With at least 2 household contacts remaining in home quarantine at the same address
* Household contacts For each index case, the study will seek to recruit as many household contacts as possible in the same house as the index case. All household contacts of the index case remaining in home quarantine in the same house as the index case will be asked to participate.

Exclusion Criteria:

* Covid-19 patients with a negative indication for home isolation, or having less than 2 household contacts remaining in home quarantine at the same address. For fingerprick blood collection, participants who have a medical indication against fingerprick blood collection will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: laboratory confirmed Sars-Cov-2 cases and their household contacts.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2020-03-26 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2020-05-13 (Actual)

PRIMARY OUTCOMES:
Mucosal antibodies | Day 0
  Descriptive analysis of SARS-CoV-2 IgG, IgM and IgA concentrations in nasal fluid
Mucosal antibodies | Day 3 (index cases)
  Descriptive analysis of SARS-CoV-2 IgG, IgM and IgA concentrations in nasal fluid
Mucosal antibodies | Day 6 (index cases)
  Descriptive analysis of SARS-CoV-2 IgG, IgM and IgA concentrations in nasal fluid
Mucosal antibodies | Day 7 (household contacts)
  Descriptive analysis of SARS-CoV-2 IgG, IgM and IgA concentrations in nasal fluid
Mucosal antibodies | Day 14 (household contacts)
  Descriptive analysis of SARS-CoV-2 IgG, IgM and IgA concentrations in nasal fluid
Mucosal antibodies in all participants | Day 28
  Descriptive analysis of SARS-CoV-2 IgG, IgM and IgA concentrations in nasal fluid

SECONDARY OUTCOMES:
SARS-CoV-2 infection | day 0
  SARS-CoV-2 PCR on nasopharyngeal swab and throat swab
Serum antibodies | day 28
  Descriptive analysis of SARS-CoV-2 antibody concentrations in serum at day 28.
Functional antibody assays | Day 0
  Descriptive analysis of the functionality of SARS-CoV-2 mucosal and serum antibodies
Functional antibody assays | Day 3 (index cases)
  Descriptive analysis of the functionality of SARS-CoV-2 mucosal and serum antibodies
Functional antibody assays | Day 6 (index cases)
  Descriptive analysis of the functionality of SARS-CoV-2 mucosal and serum antibodies
Functional antibody assays | Day 7 (household contacts)
  Descriptive analysis of the functionality of SARS-CoV-2 mucosal and serum antibodies
Functional antibody assays | Day 14 (household contacts)
  Descriptive analysis of the functionality of SARS-CoV-2 mucosal and serum antibodies
Functional antibody assays | Day 28
  Descriptive analysis of the functionality of SARS-CoV-2 mucosal and serum antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Diavatopoulos, Dr, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Froberg J, Koomen VJCH, van der Gaast-de Jongh CE, Philipsen R, GeurtsvanKessel CH, de Vries RD, Baas MC, van der Molen RG, de Jonge MI, Hilbrands LB, Huynen MA, Diavatopoulos DA. Primary Exposure to SARS-CoV-2 via Infection or Vaccination Determines Mucosal Antibody-Dependent ACE2 Binding Inhibition. J Infect Dis. 2024 Jan 12;229(1):137-146. doi: 10.1093/infdis/jiad385. PMID 37675756